CLINICAL TRIAL: NCT04103879
Title: A Phase II Open-Label Study of UM171-Expanded Cord Blood Transplantation in Patients With High and Very High Risk Acute Leukemia/Myelodysplasia
Brief Title: US Study of UM171-Expanded CB in Patients With High Risk Leukemia/Myelodysplasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ExCellThera inc. (Industry)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001-CB.004; Study 8743 (Other: FHCRC)
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: High Risk Hematological Malignancy; Cord Blood Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ECT-001-Expanded CB (Experimental): Patients will receive a myeloablative conditioning regimen.
  The cord to be expanded will undergo CD34+ selection. The CD34- product is cryopreserved and will be thawed and infused on Day +1 post-transplant. The CD34+ product will be placed in a closed culture with UM171 for a 7-day expansion and is infused on Day 0.
  Patients will receive standard supportive care and GVHD prophylaxis (such as MMF and tacrolimus).
  Interventions: Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant)

INTERVENTIONS:
Biological: ECT-001-CB (UM171-Expanded Cord Blood Transplant) — Conditioning: High dose TBI (1320 cGy TBI + Fludarabine 75 mg/m2 + Cyclophosphamide 120 mg/kg) or Intermediate Intensity regimen (400 cGy TBI + Fludarabine 150 mg/m2 + Cyclophosphamide 50 mg/kg + Thiotepa 10 mg/kg).
  Single UM171-Expanded CB transplant (CD34+: 2.5-50x10E5/kg, CD3+>1x10E6/kg)
  Immunosuppression: Tacrolimus/MMF

SUMMARY:
Cord blood (CB) transplants are an option for patients lacking an HLA identical donor but are hampered by low cell dose, prolonged aplasia and high transplant related mortality. UM171, a novel and potent agonist of hematopoietic stem cell self renewal could solve this major limitation, allowing for CB's important qualities as lower risk of chronic GVHD and relapse to prevail. In a previous trial (NCT02668315), the CB expansion protocol using the ECT-001-CB technology (UM171 molecule) has proven to be technically feasible and safe. UM171 expanded CB was associated with a median neutrophil recovery at day (D)+18 post transplant. Amongst 22 patients who received a single UM171 CB transplant with a median follow-up of 18 months, risk of TRM (5%) and grade 3-4 acute GVHD (10%) were low. There was no moderate-severe chronic GVHD. Thus, overall and progression free survival at 12 months were impressive at 90% and 74%, respectively. The UM171 expansion protocol allowed access to smaller, better HLA matched CBs as >80% of patients received a 6-7/8 HLA matched CB. Interestingly there were patients with high-risk hematologic malignancies and multiple comorbidities (5 patients who had already failed an allogeneic transplant and 5 patients with refractory/relapsed acute leukemia/aggressive lymphoma). Despite this high risk population, progression was 20% at 12 months.

This new study seeks to test a similar strategy in a group of patients with high risk acute leukemia/myelodysplasia.

ELIGIBILITY:
Inclusion Criteria:

1. High and very high-risk hematologic malignancy defined as:

   1. Acute Myeloid Leukemia (Primary induction failure, Chemorefractory relapse, Relapse after allogeneic or autologous transplant, High risk AML in CR1, ≥ CR2)
   2. Acute Lymphoid leukemia (Primary induction failure, High risk ALL in CR1, ≥ CR2, Chemorefractory relapse, Relapse after allogeneic or autologous transplant)
   3. Myelodysplastic syndrome (Relapse after allogeneic or autologous transplant, ≥10% blasts within 30 days of start of conditioning regimen, Poor and very poor cytogenetics abnormalities, CMML with HCT-specific CPSS score high or intermediate-2, Stable disease, Progressive disease while on azacitidine).
   4. Chronic myelogenous leukemia (Patients who progressed to blast crisis)
2. Availability of 2 CBs ≥ 4/6 HLA match with pre-freeze CD34+ cell count ≥0.5 x 10E5/kg and TNC≥1.5 x 10E7/kg
3. Karnofsky ≥70.
4. LVE fraction ≥ 40% or fractional shortening >22%
5. FVC, FEV1 and DLCOc ≥ 50% of predicted
6. Bilirubin < 2 x ULN; AST and ALT ≤ 2.5 x ULN; alkaline phosphatase ≤ 5 x ULN.
7. Creatinine < 2.0 mg/dl.
8. HCT-CI ≤3 if patients have ≥5% blasts in the bone marrow and HCT-CI ≤5 if 60-65 years old.

Exclusion Criteria:

1. Allogeneic myeloablative transplant within 6 months.
2. Autologous hematopoietic stem cell transplant within 6 months.
3. Active or recent invasive fungal infection.
4. Presence of a malignancy other than the one for which the UCB transplant is being performed and the expected survival related to the malignancy is estimated to be less than 75% at 5 years.
5. HIV positivity.
6. Hepatitis B or C infection with measurable viral load.
7. Liver cirrhosis.
8. Pregnancy, breastfeeding or unwillingness to use appropriate contraception.
9. Any abnormal condition or laboratory result that is considered by the principal investigator capable of altering patient condition or study outcome.
10. Active central nervous system involvement.
11. Chloroma > 2 cm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events of ECT-001-CB | 100 days post-transplant
  All AEs will be graded in severity according to the modified (for HSCT) CTCAE (v. 5.0)
Adverse events of ECT-001-CB | 2 years post-transplant
  All AEs will be graded in severity according to the modified (for HSCT) CTCAE (v. 5.0)
Relapse-free survival | At 1-year post-transplant
  RFS will be measured from time of transplant until disease relapse, death or last follow-up
Relapse-free survival | At 2-year post-transplant
  RFS will be measured from time of transplant until disease relapse, death or last follow-up

SECONDARY OUTCOMES:
Time to Neutrophil and Platelet engraftment | First 60 days
  Neutrophil engraftment (the first day of attainment of an absolute neutrophil count ≥0.5 x 10E9/L for 3 consecutive days. Time to ANC ≥ 0.1 x 10E9/L will also be documented) and platelet engraftment (first day of a sustained platelet count ≥ 20 x 10E9/L with no platelet transfusion in the preceding 7 days)
Incidence of transplant related mortality | At day 100 post-transplant
  TRM is defined as any death of any cause other than malignant relapse, occurring after the commencement of conditioning regimen that could be related to the transplantation procedure
Incidence of transplant related mortality | At 1-year post-transplant
  TRM is defined as any death of any cause other than malignant relapse, occurring after the commencement of conditioning regimen that could be related to the transplantation procedure
Incidence of GVHD | At 2 years post-transplant
  Acute and chronic GVHD by NIH criteria
Incidence of grade 3 or higher infectious complications | At 2 years post-transplant
  Any of infections requiring systemic therapy, e.g., invasive candidiasis, aspergillus, other invasive fungi, CMV, adenovirus, EBV, HHV-6, HSV, VZV, PCP, toxoplasmosis and mycobacterium
Incidence of pre-engraftment/engraftment syndrome requiring therapy | At 2 years post-transplant
GRFS and CRFS | At 1-year post-transplant
  GRFS and CRFS will be measured from time of transplant until disease relapse, death or last follow-up
GRFS and CRFS | At 2-year post-transplant
  GRFS and CRFS will be measured from time of transplant until disease relapse, death or last follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Colorado School of Medicine. Anschutz Medical Campus, Aurora, Colorado
  - Fred Hutchinson / University of Washington Cancer Consortium, Seattle, Washington
- Erasmus Medical Center, Rotterdam, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR